CLINICAL TRIAL: NCT04611750
Title: Pharmacological Intervention for Symptomatic Mild Sleep Disordered Breathing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Apnimed (Industry)
Responsible Party: Principal Investigator, Scott Aaron Sands, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002259
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sleep Disordered Breathing
Keywords: Inspiratory flow limitation; Snoring; Mild Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Medication (AD036) (Experimental): Participants will take AD036 QHS for 14 days.
  Interventions: Drug: AD036
- Placebo Medication (Placebo Comparator): Participants will take placebo QHS for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD036 — AD036 will be given for 14 days
  Arms: Active Medication (AD036)
Drug: Placebo — Placebo will be given for 14 days
  Arms: Placebo Medication

SUMMARY:
Currently, there is no pharmacological intervention for mild symptomatic obstructive sleep disordered breathing (SDB) in the form of loud habitual snoring, inspiratory flow limitation (i.e. upper airway resistance syndrome), or mild sleep apnea. Here the investigators study the effect on SDB of stimulating pharyngeal muscles during sleep with AD036. The key hypothesis of the study is that AD036 is superior to placebo on self-reported and objective measures of SDB severity.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled 2-period crossover study. Each crossover period will consist of 14 days of QHS dosing of either AD036 or placebo, with a washout period of 7 days between each period.

Polysomnography will be performed at screening (baseline) and on the last dosing day of each of the two crossover dosing period.

The trial will enroll participants until a total of 24 responders are randomized into the crossover portion of the study.

ELIGIBILITY:
Inclusion Criteria at Enrollment:

* Between 25 to 70 years of age, inclusive
* SRQ at screening ≥ 4 (at least mild impact of snoring)
* ESS at screening ≤ 12 (absence of sleepiness)
* BMI between 18.5 and 40 kg/m2, inclusive.
* Use of specified contraceptive methods if appropriate

Inclusion Criteria for First Study Phase (Run-in Period):

* AHI ≥5-10, or AHI 0-<5 if either:
* Snoring frequency (100dB snoring for >10% of sleep) by tracheal microphone, or
* Flow limitation frequency (>50% obstruction for >10% of sleep).
* PGI-S that improves by at least 1 point during AD036 run-in period

Inclusion Criteria for Randomization:

• PGI-S that improves by at least 1 point during AD036 run-in period.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* History of narcolepsy
* Clinically significant craniofacial malformation
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control.
* Clinically significant neurological disorder, including epilepsy/convulsions.
* History of schizophrenia, schizoaffective disorder or bipolar disorder
* History of attempted suicide or suicidal ideation within 1 year prior to screening, or current suicidal ideation.
* History of clinically significant constipation, gastric retention, or urinary retention.
* Positive screen for drugs of abuse or substance use disorder
* A significant illness or infection requiring medical treatment in the past 30 days.
* Clinically significant cognitive dysfunction.
* Untreated narrow angle glaucoma.
* Women who are pregnant or nursing.
* History of using oral or nasal devices for the treatment of OSA or snoring; may enroll as long as the devices are not used during participation in the study.
* History of using devices to affect participant sleeping position for the treatment of OSA or snoring, e.g. to discourage supine sleeping position; may enroll as long as the devices are not used during participation in the study.
* History of oxygen therapy (last 12 months).
* Use of medications from the list of disallowed concomitant medications during study participation.

  * MAOIs or other drugs that affect monoamine concentrations (e.g., rasagiline) [MAOIs are contraindicated for use with atomoxetine]
  * Selective Serotonin Reuptake Inhibitors (e.g., paroxetine)
  * Selective Norepinephrine Reuptake Inhibitors (e.g., duloxetine)
  * Norepinephrine Reuptake Inhibitors (e.g., reboxetine)
  * Alpha-1 antagonists (e.g., tamsulosin)
  * Tricyclic antidepressants (e.g., desipramine)
  * Centrally acting antihypertensives (e.g. clonidine, alpha-methyl-DOPA)
  * CYP2D6 inhibitors
  * Strong CYP3A4 inhibitors (e.g., ketoconazole)
  * Benzodiazepines and other anxiolytics or sedatives
  * Nonbenzodiazepine hypnotics
  * Opioids
  * Muscle relaxants
  * Pressor agents
  * Drugs with clinically significant cardiac QT-interval prolonging effects
  * Drugs known to lower seizure threshold (e.g., chloroquine)
  * Amphetamines
  * Antiepileptics
  * Antiemetics
  * Modafinil or armodafinil
  * Beta2 agonists, (e.g., albuterol)
  * Antipsychotics
  * Anticholinergics and anticholinesterase inhibitors, including drugs with substantial anticholinergic side effects, (e.g., first generation antihistamines)
  * Sedating antihistamines
  * Pseudoephedrine, phenylephrine, oxymetazoline
  * Nicotine replacement products
  * Most drugs for Parkinson's, Alzheimer's, Huntington's, Amyotrophic Lateral Sclerosis, or drugs for other neurodegenerative diseases
* Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, strong cytochrome P450 2D6 (CYP2D6) inhibitors, or monoamine oxidase inhibitors (MAOI) within 14 days of the start of treatment, or concomitant with treatment.
* Use of another investigational agent within 30 days or 5 half-lives prior to dosing, whichever is longer.
* <5 hours typical sleep duration.
* Smoking more than 10 cigarettes or 2 cigars per day.
* Unwilling to use specified contraception.
* Unwilling to limit alcohol consumption to no greater than 2 units/day or less for men, or 1 unit/day for women, not to be consumed within 3 hours of bedtime.
* Unwilling to limit caffeinated beverage intake (e.g., coffee, cola, tea) to 400 mg/day or less of caffeine (approximately 4 cups of coffee); caffeine not to be used within 3 hours of bedtime.
* Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
* Participant considered by the investigator, for any reason, an unsuitable candidate to receive AD036 or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Snoring Relationship Questionnaire (SRQ) | 14 days
  Self-reported impact of snoring on relationship and quality of life for patients and bedpartners, 0-20 scale, 0 lowest severity, 20 highest severity

SECONDARY OUTCOMES:
Snoring Frequency | 14 days
  Snoring frequency, % breaths during sleep >100dB by tracheal microphone
Flow Limitation Frequency | 14 days
  Flow limitation frequency, % breaths during sleep >50% obstructed per airflow shape (Mann D et al ERJ)
Apnea-Hypopnea Index | 14 days
  Apnea-Hypopnea Index, events/hr (hypopneas per 4% desaturation)

OTHER OUTCOMES:
Snoring Intensity | 14 days
  Mean tracheal sound pressure, presented in dB
Flow Limitation Severity, % | 14 days
  Median overnight flow limitation severity (Mann et al ERJ) in %, 0% is maximal flow limitation, 100% is absence of flow limitation
Hypoxic Burden | 14 days
  Area under curve of pulse oxygen saturation due to respiratory events (Azarbarzin et al EHJ method) in %desaturation.min/hr
Sleep Apnea Quality of Life Index (Short) | 14 days
  Sleep-related quality of life on 1-7 scale, 1 is lowest quality of life, 7 is highest quality of life
Snoring Self-Evaluation Survey (SSES) | 14 days
  Snoring-related symptoms and quality of life for the snorer on a 0-16 scale, 0 represents absence of snoring and related symptoms, 16 represents maximal snoring and related symptoms
Snoring Bedpartner-Evaluation Survey (SBES) | 14 days
  Snoring-related quality of life for the bedpartneron a 0-16 scale, 0 represents absence of snoring and related symptoms, 16 represents maximal snoring and related symptoms
Epworth Sleepiness Scale | 14 days
  Sleepiness 0-24 scale, 0 least sleepy, 24 most sleepy
Visual Analog Scale for Treatment Satisfaction | 14 days
  Treatment Satisfaction 0-10 scale, 0 most dissatisfied, 5 neutral, 10 most satisfied
Participant Global Impression of Severity (PGI-S) of SDB symptoms | 14 days
  Self-reported Symptom Severity 0-4 scale, 0 lowest severity, 4 highest severity

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital; Bradley A Edwards, PhD, Principal Investigator — Monash University
Locations (2):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- Monash University, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
We plan not to share data

REFERENCES:
- [Derived] Hynes DJ, Mann DL, Landry SA, Joosten SA, Edwards BA, Hamilton GS. Night-to-night variability in obstructive sleep apnea severity, the physiological endotypes, and the frequency of flow limitation. Sleep. 2025 Apr 11;48(4):zsae295. doi: 10.1093/sleep/zsae295. PMID 39688178